CLINICAL TRIAL: NCT07267598
Title: Evaluating the Effectiveness of a 26 °C Indoor Temperature Limit to Mitigate Physiological Strain in Young, Habitually Active Adults
Brief Title: Suitability of a 26 °C Indoor Environment for Mitigating Heat Strain in Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Professor and University Research Chair, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2025-10B
Record Dates: First submitted 2025-11-21; First posted 2025-12-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Heat Stress; Physiological Stress; Cognitive Change
Keywords: Indoor overheating; Indoor temperatures; Heat wave; Thermoregulation; Heat strain; Heat vulnerability; Hyperthermia; Thermal comfort; Activities of daily living; Clothing insulation
MeSH Terms: conditions — Heat Stress Disorders; Hyperthermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to indoor temperature upper limit without physical activity and added clothing. (Experimental): Participants, dressed in light clothing (t-shirt, shorts and socks), perform seated rest while exposed daylong (8 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated indoor temperature upper limit
- Exposure to indoor temperature upper limit with physical activity and added clothing. (Experimental): Participants, dressed in light clothing (t-shirt, shorts and socks) and an added clothing layer (sweatshirt and sweatpants), perform light exercise (i.e., stepping, representing activities of daily living, 4-4.5 METS) every hour (with exception of lunch hour) while exposed daylong (8 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated indoor temperature upper limit

INTERVENTIONS:
Other: Simulated indoor temperature upper limit — Young adults exposed to an 8-hour simulated exposure.

SUMMARY:
While an indoor upper temperature limit of 26 °C has been shown to protect heat-vulnerable older adults (DOI: 10.1289/EHP11651), this guideline has not been verified in young, habitually active adults. Public health recommendations during hot weather typically emphasize staying in cool environments, avoiding strenuous activity, wearing lightweight clothing, and maintaining adequate hydration. However, young adults may be less likely to follow these guidelines. They often do not reduce their physical activity during extreme heat events and may overdress for fashion, cultural, or religious reasons. These behaviors can impose an additional thermoregulatory burden and lead to greater physiological strain during heat exposure, even though young adults generally have a higher capacity for heat dissipation than older individuals. Accordingly, it is important to evaluate whether an indoor temperature limit of 26 °C is sufficient to protect young, habitually active adults.

To address this gap, the investigators aim to assess changes in body temperature and cardiovascular strain in young, habitually active adults (18-29 years) during an 8-hour exposure to the recommended indoor upper temperature limit of 26 °C and 45% relative humidity (humidex of 29, considered comfortable). Participants will complete two conditions:

A) seated rest while dressed in light clothing (T-shirt, shorts, and socks), and B) light exercise (stepping to simulate activities of daily living, 4-4.5 METs) performed once per hour (except for the lunch hour) while dressed in light clothing plus an additional insulating layer (sweatshirt and sweatpants).

This experimental design will allow investigators to determine the effects of added clothing insulation and light activity-representative of typical daily behaviors-on physiological strain in young adults, and to assess whether refinements to the recommended 26 °C indoor temperature limit are warranted for this population.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.
* Healthy young adults without chronic disease (e.g., type 1 diabetes, hypertension)

Exclusion Criteria:

* Endurance trained (i.e., engaged in regular physical training activities more than 3 times a week for more than 1 hour per session).
* Undergoing passive heat exposures such as regular of saunas, warm-water immersion, other.
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable.
* Current pregnancy

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-13 (Estimated)

PRIMARY OUTCOMES:
Core temperature (Peak) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the 8 hour exposure to the simulated indoor temperature upper limit.
Core temperature (AUC) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Areas under the curve (AUC) of rectal temperature during the 8 hour exposure to the simulate indoor temperature upper limit.
Core temperature end of daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Rectal temperature measured at hour 8 of exposure to indoor temperature limit (15-min average).
Mean skin temperature (Peak) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Peak mean skin temperature (15 min average) during exposure. Mean skin temperature as calculated from skin temperature measured across 7 body regions is measured continuously throughout the 8 hour exposure to the simulated indoor temperature upper limit.
Mean skin temperature (AUC) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Areas under the curve (AUC) of mean skin temperature as calculated over 7 body regions during the 8 hour exposure to the simulate indoor temperature upper limit.
Mean skin temperature end of daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Mean skin temperature measured over 7 body regions at hour 8 of exposure to indoor temperature limit (15-min average).
Heat rate (Peak) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Peak heart rate (15 min average) during exposure. Heart rate is measured continuously throughout the 8 hour exposure to the simulated indoor temperature upper limit.
Heart rate (AUC) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Areas under the curve (AUC) of heart rate during the 8 hour exposure to the simulate indoor temperature upper limit.
Heart rate end of daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Heart rate measured at hour 8 of exposure to indoor temperature limit (15-min average).
Heart rate variability: RMSSD during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the supine position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of supine rest).
Heart rate variability: SDNN during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the supine position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of supine rest).
Cardiac response to standing from supine (30:15 ratio) during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Cardiac response to standing evaluated as the ratio between the highest R-wave to R-wave interval (lowest heart rate) measured at the 30th heart beat after standing from supine (+/- 5 beats) and the lowest R-wave to R-wave interval (highest heart rate) measured at the 15th heart beat after standing (+/- 5 beats). Cardiac response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic response to standing from supine during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic blood pressure during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures).
Diastolic blood pressure during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures).
Rate pressure product during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Rate pressure product, an index of myocardial work and strain, calculated as systolic blood pressure x heart rate.
Reaction time during daylong exposure to indoor temperature limit (cognitive function). | At the start (hour 0) and end of 8 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of reaction time. Participants will be asked to initiate a movement of the device in response to a visual cue.
Impulse control during daylong exposure to indoor temperature limit (cognitive function). | At the start (hour 0) and end of 8 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of impulse control. Participants will be asked to respond to both "go" and "no-go" visual cues. In response to the "go" cue, participants will initiate a movement of the device.
CDC 4-Stage Balance Test during daylong exposure to indoor temperature limit (postural stability). | At the start (hour 0) and end of 8 hour daylong exposure
  To assess postural stability, participants hold a tablet to their chest, then auditory cues guide participants through four consecutive stances, feet side by side, instep of one foot touching the big toe of the other foot, tandem stand with one foot in front of the other, heel touching toe, and stand on one foot. The balance assessment will be evaluated based on movement detected by an accelerometer integrated into the hardware of the tablet device (Sway Medical Inc).
BTrackS Balance Assessment during daylong exposure to indoor temperature limit (postural stability). | At the start (hour 0) and end of 8 hour daylong exposure
  To assess postural stability, participants will be asked to stand on a BTracks force plate with their feet spread out to shoulder width while looking straight ahead. The assessment will comprise of one trial lasting 120 seconds in length. Center of pressure (COP) vector data along vertical (y) and horizontal (x) axes will be summed for the total path excursion length (cm) during each trial.
Fluid consumption during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Fluid loss during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for food consumption).
Change in plasma volume during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Change in plasma volume from baseline values calculated from duplicate measurements of hemoglobin and hematocrit at the start and end of each exposure using the technique by Dill and Costill.
Thermal comfort scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") ranging from "very uncomfortable" to "comfortable".
Thirst sensation scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Thirst sensation assessed via a visual analog scale ranging from "very, very thirsty" to "not thirsty at all".
Arousal scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Felt arousal scale assessed via a visual analog scale ("How worked up are you?") ranging from "high arousal" to "low arousal".
Thermal sensation scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Thermal sensation assessed via a visual analog scale ("How hot do you feel?") ranging from "extremely hot" to "neutral"(midpoint: hot)
Thermal sensation 2 scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Thermal sensation assessed via a visual analog scale ("How do you feel?") ranging from "hot" to "cold"(midpoint: neutral)
Orthostatic intolerance symptoms assessment during daylong exposure to indoor temperature limit. | At end of 8 hour daylong exposure
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance during the lying to standing tests. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort".
Feel good scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Feel good assessed via a visual analog scale ("How good do you feel?") ranging from "very good" to "very bad"(midpoint: neutral).
Perceived exertion scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Perceived exertional assessed via a visual analog scale ("How hard are you working?") ranging from "no exertional at all" to "maximal exertion".
Hydration status during daylong exposure to indoor overheating | At the start (hour 0) and end of 8 hour daylong exposure
  Hydration status measured via assessing the urine specific gravity of a urine sample.
Activity levels during daylong exposure to indoor overheating | End of 8 hour daylong exposure
  Activity levels assessed via a wearable monitor (Actical) containing an accelerometer worn on the wrist and hip.

SECONDARY OUTCOMES:
Profiles of Mood States (POMS) during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives. For each individual item, participants were asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) were summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure [24, 25].
  Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score was calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").
Sleep quality and quantify assessment during daylong exposure to indoor temperature limit. | At the start of 8 hour daylong exposure.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that works by asking 19 questions about a person's sleep habits over the past month. It is scored by evaluating seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored from 0 to 3, and these are summed to create a global score from 0 to 21, where a higher score indicates poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada